CLINICAL TRIAL: NCT01620996
Title: A Novel Approach to Cardiovascular Health by Optimizing Risk Management (ANCHOR): A Primary Prevention Initiative Examining The Impact Of Global Risk Factor Assessment & Management On Health Care In Nova Scotia
Brief Title: A Novel Approach to Cardiovascular Health by Optimizing Risk Management (ANCHOR)
Acronym: ANCHOR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Collaborators: Cape Breton District Health Authority (Unknown); Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: CD-2005-267
Record Dates: First submitted 2012-06-13; First posted 2012-06-15 (Estimated); Last update posted 2022-11-15 (Actual); Status verified 2008-06

CONDITIONS: Cardiovascular Risk Reduction of Having a Coronary Event
Keywords: preintervention and postintervention cohort longitudinal prospective study
MeSH Terms: interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Active Comparator): Duffus Street Medical Centre
  Interventions: Behavioral: Minimal Intervention; Behavioral: Motivational Interviewing; Behavioral: Motivational Enhancement
- 2 (Active Comparator): Sydney Family Practice
  Interventions: Behavioral: Minimal Intervention; Behavioral: Motivational Interviewing; Behavioral: Motivational Enhancement
- no counseling (No Intervention): HRA assessment pre and post but no counselling

INTERVENTIONS:
Behavioral: Minimal Intervention — There is no clear definition of this term and it has been used by many different groups to refer to attempts to alter behavior by providing very brief, focused interventions. A slightly more developed model guiding intervention is called the 5-A model. This refers to the acronym Ask, Advise, Assess, Assist and Arrange. This model has been endorsed by the US Public Health Department, who has incorporated the 5-A approach into their clinical practice guidelines (A Clinical Practice Guideline for Treating Tobacco Use and Dependence; A US Public Health Service Report. JAMA, June 20, 2000 - Vol 283 No. 24; see also http://www.surgeongeneral.gov/tobacco/tobaqrg.htm).
  Arms: 1; 2
Behavioral: Motivational Interviewing — Motivational Interviewing has its roots in alcohol abuse counseling and was pioneered by Miller and Rollnick. It is an approach to counseling that is geared toward increasing an individual's motivation, or buy-in, to the work that needs to be done to reduce substance dependence. Miller and Rollnick offer the approach as a brief intervention (hence some confusion with the term minimal intervention) guided by the following mediators of change, which they call ingredients of change, summarized by the Acronym FRAMES:
  FEEDBACK of personal risk or impairment Emphasis on personal RESPONSIBILITY for change Clear ADVICE to change A MENU of alternative change options Therapist EMPATHY Facilitation of client SELF-EFFICACY or optimism
  These mediators/ingredients are delivered by the clinician using the following principles:
  Express Empathy Develop Discrepancy Avoid Argumentation Roll with Resistance Support Self-Efficacy
  Arms: 1; 2
Behavioral: Motivational Enhancement — Motivational enhancement is the most comprehensive term and reflects the integration of two major theorists; Millner and Rollnick on the one hand, and Prochaska and his colleagues on the other. The work of Miller and Rollnick occurred within substance abuse, primarily alcohol abuse and is best summarized in the section above on motivational interviewing. As Prochaska's work, which initially began in the area of smoking cessation but quickly expanded to include wide-ranging health behaviours, developed Miller and Rollnick incorporated his work with theirs.Prochaska's model derives from his long term study of the process of behaviour change regardless of the model of intervention implemented.The model is often referred to as the stages of change model, or readiness to change model.
  The stages of change model identifies five separate stages; precontemplation,contemplation, preparation, action, and maintenance
  These stages are specific to different behaviours.
  Arms: 1; 2

SUMMARY:
Study Purpose and Design

The goal of this study is to improve CVD risk in a primary care adult population, with the following primary objectives

1. To improve management of global cardiovascular risk of patients within two primary care practices, thereby improving their overall cardiac health.
2. To increase patient compliance with lifestyle aimed at pharmaceutical interventions aimed at decreasing global cardiovascular risk.

Secondary objectives of the study are:

1. To examine the utility of a process to improve the management of global cardiovascular risk of patients within two primary care practices.
2. To explore the utility of a process that links primary care practices with existing community resources in order to manage cardiac risk factors better among individuals within those primary care practices.
3. To determine the economic impact of a global risk assessment and management process within a primary care setting.

DETAILED DESCRIPTION:
The Burden of Cardiovascular Disease

Cardiovascular disease (CVD) remains the major cause of mortality in the developed world, accounting for almost 40% of all deaths in both the United States and Canada. It represents a substantial financial drain on society and contributes a significant burden to health care systems that are already under strain. Major modifiable risk factors for CVD include elevated blood pressure, cigarette smoking, elevated total plasma cholesterol and low high-density lipoproteins, diabetes, obesity, and sedentary lifestyle, at least one of which is present in 80% of Canadians. Circulatory diseases (particularly heart disease, stroke and hypertension) cost the Nova Scotia health care system an estimated $961 million dollars per year. In Nova Scotia cardiovascular disease kills an estimated 2,900 Nova Scotians every year accounting for nearly 36% of all deaths in the province.

Cardiovascular Disease Prevention in Primary Care Settings

There is strong evidence linking improved risk factors among populations to improved health outcomes, and both epidemiological and community research have illustrated that the bulk of non-communicable diseases (NCDs) such as CVD are preventable, or at least their occurrence can be postponed. Because primary care physicians are most often the first point of contact for individuals in need of health care, general practice is well placed to facilitate change in patients' risk factor status and ensure more effective treatment of risk factors such as hypertension and hyperlipidemia. Currently primary care service delivery is expanding to include a broader network of providers such as nurses, dieticians, and pharmacists to enable more effective risk factor identification and management, and health promotion and disease prevention efforts across the continuum of care.

Nova Scotia Context

Currently in Nova Scotia, population health and disease prevention initiatives are underway that will support and reinforce the work of the current study, including primary health care transition fund initiatives, and strategic directions from the Office of Health Promotion that address major risk factors for cardiovascular disease. These provincial initiatives together with local projects ongoing in several communities provide an ideal opportunity for interfacing with a primary care global risk reduction initiative.

Study Purpose and Design

The goal of this study is to improve CVD risk in a primary care adult population, with the following primary objectives

1. To improve management of global cardiovascular risk of patients within two primary care practices, thereby improving their overall cardiac health.
2. To increase patient compliance with lifestyle and pharmaceutical interventions aimed at decreasing global cardiovascular risk.

Secondary objectives of the study are:

1. To examine the utility of a process to improve the management of global cardiovascular risk of patients within two primary care practices.
2. To explore the utility of a process that links primary care practices with existing community resources in order to manage cardiac risk factors better among individuals within those primary care practices.
3. To determine the economic impact of a global risk assessment and management process within a primary care setting.

The intervention will be led by a study coordinator in each primary care setting and consist of a recruitment strategy, global risk factor assessment, behaviour change counseling, and risk factor management strategies based on the 5A's framework (assess, advise, agree, assist and arrange follow-up). Supports will be provided to study participants in making behaviour changes including counseling and follow-up, behaviour change tools, print resources, group education sessions, and an inventory of and links to community programs. Medication reviews and physician referrals will also be completed as required.

A Steering Committee will guide the project and includes membership from the Principal Investigators, representatives from Pfizer Canada, Capital District Health Authority, the Cape Breton District Health Authority and the Nova Scotia Department of Health; and community stakeholders including community pharmacy, a physician and/or nurse from each site, other relevant allied health professionals (e.g., nutritionist) and the CEO from the Heart and Stroke Foundation of Nova Scotia. The initiative will be conducted over a three-year period and will comprise three phases as outlined in the following table.

Research Methodology

This is a pre-intervention and post-intervention longitudinal, prospective pilot study to evaluate study participants achievement of CVD risk factor reduction. The research will include a combination of quantitative and qualitative data to judge effectiveness of the interventions and to describe the intervention as it is implemented. The effectiveness of the approach will be examined using pre and post measures of key outcome variables. In addition to these outcome measures, process evaluation will monitor and assess the implementation of the interventions. The study will include baselines measurement, periodic assessments of process measures, outcome measurement and follow-up measurement. Following the baseline measurement through the GRA, patients will receive risk management interventions.

The data will be analyzed using both quantitative and qualitative methods. Pre and post outcome measures will be analyzed using descriptive analytical techniques comparing means for continuous measures and proportions for categorical measures. Qualitative data will be managed and analyzed either manually or via QSR NUD*IST (Qualitative Solutions and Research Non-numerical Unstructured Data Indexing Searching and Theory-building) software. The qualitative analysis will consist of both content and thematic analysis.

Sustainability and Dissemination

The project will involve collaboration and integration with primary health care renewal efforts and community resources to build on existing infrastructure and thereby help to facilitate sustainability. Capacity building within primary care settings and mobilization of existing resources will also help to ensure a sustainable resource. Steering Committee members and other partners will ensure the project results and products are shared with their organizations and networks, and also more widely across the province. Project findings will be published in appropriate peer reviewed publications to further share the learning and disseminate findings.

ELIGIBILITY:
Inclusion Criteria:

* 30 years of age
* a patient of the primary care practices involved in the study
* able to provide informed consent

Exclusion Criteria:

* under the age of 30
* not a patient of the primary care practices
* unable to provide informed consent

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1708 (Actual)
Dates: Start 2006-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
achievement of targeted mean reductions in overal global risk within patient risk strata Proportion of patients achieving their targeted mean reduction in global risk within risk strata | 12 months

SECONDARY OUTCOMES:
determine the economic impact of a global risk assessment management process within a primary care setting | 12 months
percentage of patients that reduced at least one risk category from baseline | 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Duffus Health Centre, Halifax, Nova Scotia, Canada

REFERENCES:
- [Derived] Cox JL, Vallis TM, Pfammatter A, Szpilfogel C, Carr B, O'Neill BJ. A novel approach to cardiovascular health by optimizing risk management (ANCHOR): behavioural modification in primary care effectively reduces global risk. Can J Cardiol. 2013 Nov;29(11):1400-7. doi: 10.1016/j.cjca.2013.03.007. Epub 2013 Jun 21. PMID 23796526